CLINICAL TRIAL: NCT02179229
Title: Effect of Pre- and Probiotics on P-cresol Plasma Levels in Patients Bearing a Kidney Allograft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Bruna Guida, M.D., Federico II University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Syn-Graft Study
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Kidney transplantation; pCresol; Immunosuppressant drugs
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONTROL (Placebo Comparator): Patient in the CONTROL arm will receive a powder containing only tapioca-resistant starch comparable in colour, texture and taste to the synbiotic.
  Interventions: Dietary Supplement: CONTROL
- SYNBIOTIC (Experimental): Patients in this group will receive Probinul neutro® a synbiotic preparation containing (perpacket): lyophilised bacteria (5×109 Lactobacillus plantarum, 2×109 Lactobacillus casei subsp. rhamnosus and 2×109 Lactobacillus gasseri, 1×109 Bifidobacterium infantis and 1×109 Bifidobacterium longum, 1×109 Lactobacillus acidophilus, 1×109 Lactobacillus salivarius and 1×109 Lactobacillus sporogenes and 5×109 Streptococcus thermophilus), prebiotic inulin (2.2 g; VB Beneo Synergy 1) and 1.3 g of tapioca-resistant starch.
  Interventions: Dietary Supplement: SYNBIOTIC

INTERVENTIONS:
Dietary Supplement: CONTROL — Placebo will be taken at home for four weeks as 5 g powder packets to be dissolved in water three times a day far from meals.
  Other Names: PLACEBO
  Arms: CONTROL
Dietary Supplement: SYNBIOTIC — Probinul Neutro® will be taken at home for four weeks as 5 g powder packets to be dissolved in water three times a day far from meals.
  Other Names: Probinul Neutro®
  Arms: SYNBIOTIC

SUMMARY:
The purpose of this study is to establish whether a short treatment with the synbiotic combination Probinul neutro® may decrease the plasma concentration of the uremic toxin p-cresol in patients bearing a kidney allograft. The effect of this treatment on plasma levels of immunosuppressant drugs will be evaluated as well.

DETAILED DESCRIPTION:
Marked alterations in the gut microbiome take place in patients with chronic kidney disease (CKD) that show an overgrowth of aerobic bacteria such as Enterobacteriaceae, Halomonadaceae, Moraxellaceae, and Pseudomonadaceae and a decrease of anaerobic bacteria such as Lactobacillaceae and Prevotellaceae. These changes also occur after kidney transplantation. The dysbiotic microflora produces toxic compounds such as phenols, indoles, and amines that are absorbed through the intestinal mucosa and cause systemic toxicity. Compelling evidence showed the association of one of these compounds, p-cresol and of its main metabolite p-cresylsulfate, to cardiovascular risk and mortality in CKD. Therefore, new therapeutic strategies decreasing the generation or absorption of this uremic toxin are expected to have a favorable impact on the clinical course of the disease. In the present study, the effect of the synbiotic Probinul neutro® on p-cresol concentration in patients bearing a kidney allograft will be evaluated. Synbiotics are associations of prebiotics and probiotics. Probiotics are living microorganisms such as Bifidobacterium and Lactobacillus species that are administered to repopulate the gut with a "normal" microflora. Prebiotics are non-digestible food adjuncts that can be selectively fermented by probiotics or by normal intestinal microflora. In synbiotics the prebiotic and probiotic components synergize to restore the normal gut microflora. Indeed, the probiotic and prebiotic components of the synbiotic may both affect the gut microbiome through with different mechanisms. Probiotics contain bacteria that are part of the normal microbiome and are lowered in CKD such as anaerobes of Bifidobacterium sp. and facultative anaerobes of Lactobacillus sp. These bacterial species, unable to convert aromatic aminoacids into p-cresol, may replace by competition the p-cresol-producing bacteria of the dysbiotic microflora because of their ability to release substances toxic for the dysbiotic microflora such as the bacteriocins, and to activate innate and adaptive immunity. Prebiotics, instead, promote the growth of non-p-cresol producing commensal flora, including lactobacilli and bifidobacteria that selectively metabolize the oligosaccharides contained in prebiotic. The combined activity of pre- and probiotic is expected to reduce the production of p-cresol in the gut by decreasing the bacterial species generationg this compound. We recently showed that a short term treatment with Probinul neutro® causes, indeed, a decrease in p-cresol plasma levels in patients with satge III/IV CKD.

ELIGIBILITY:
Inclusion Criteria:

* Previous renal allograft transplantation

Exclusion Criteria:

* severe infections
* diabetes
* malignancy
* history of food intolerance
* autoimmune disorders
* severe malnutrition or clinical conditions requiring artificial feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Change in p-cresol plasma concentration | one month
  Total p-cresol (free and glucurono- or sulpho-conjugates) plasma concentration will be assessed by reverse phase HPLC at baseline, 15 and 30 days after starting synbiotic treatment.

SECONDARY OUTCOMES:
Change in bowel habits | one month
  Defecation frequency or ease, stool shape, upper or lower abdominal pain, frequency of borborygms or flatus will be assessed by asking the patients to fill a a form for the scored evaluation of GI symptoms and stool characteristics
Change in plasma immunosuppressant drug concentration | one month
  Plasma concentration of the different immunosuppressant assumed by the patient (mycophenolate mofetil, cyclosporin, tacrolimus, everolimus or sirolimus) will be assessed at baseline, 15 and 30 days after the beginning of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Bruna Guida, MD, Principal Investigator — Federico II University of Naples
Locations (1):
- Nutrition Unit of the Federico II University of Naples, Naples, Italy

REFERENCES:
- [Derived] Cooper TE, Scholes-Robertson N, Craig JC, Hawley CM, Howell M, Johnson DW, Teixeira-Pinto A, Jaure A, Wong G. Synbiotics, prebiotics and probiotics for solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 20;9(9):CD014804. doi: 10.1002/14651858.CD014804.pub2. PMID 36126902